CLINICAL TRIAL: NCT02399982
Title: Innovative Use of the Noom Monitor Mobile Application for CBT-GSH in Binge Eaters
Brief Title: Smartphone Technology and CBT-GSH in Binge Eaters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Noom Inc. (Industry); Kaiser Foundation Hospitals, Center for Health Research (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 11-0454; 5R41MH096435-02 (NIH)
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Binge Eating Disorder; Bulimia Nervosa
Keywords: Smartphone Application; mobile mental health; Binge Eating; Cognitive behavioral therapy; Eating Disorder treatment; Cognitive behavioral therapy guided self-help; self-monitoring; eating disorders; ecological momentary intervention
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia Nervosa; Bulimia; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-GSH (Active Comparator): Traditional CBT-GSH with paper and pencil self-monitoring
  Interventions: Other: CBT-GSH
- CBT-GSH + Noom Monitor (Experimental): CBT-GSH with smartphone application for self-monitoring
  Interventions: Other: CBT-GSH; Other: Noom Monitor

INTERVENTIONS:
Other: CBT-GSH — The treatment will be based on Overcoming Binge Eating. The treatment is divided into a user-friendly section on binge eating and a six-step self-help program. The first session will last 60 min, with each subsequent section lasting 20-25 minutes in length. Sessions are weekly over 3 months. Working with the therapist, participants will use the self-help guide to develop regular and moderate eating using selfmonitoring, problem solving, and other CBT techniques.
Other: Noom Monitor — This treatment will be exactly the same as CBT-GSH with the exception that all self-monitoring will be conducted through Noom Monitor and individuals will receive a specialized set of instructions on how to use the monitor. Therapists will also be asked to check feedback report on clients before each session. Therapists will receive weekly letter grades regarding each patient based on weekly level of OBEs/Purging, treatment adherence, and weekly weighing.
  Arms: CBT-GSH + Noom Monitor

SUMMARY:
This study aims to utilize emerging mobile application technology, as a tool for increasing the potency, accessibility, and efficacy of a guided self-help version of cognitive-behavioral therapy (CBT-GSH) for binge eating. The feasibility and efficacy of the adapted smartphone application created by Noom Inc., Noom Monitor, will be examined through a randomized control trial comparing CBT-GSH + APP with CBT-GSH conducted at the Mount Sinai School of Medicine's Eating and Weight Disorders Program. The investigators hypothesize that CBT-GSH with the addition of the Noom Monitor, will be significantly more acceptable, have greater uptake of self-monitoring, greater adherence to treatment, and greater reduction in objective binge episodes (OBEs) than standard CBT-GSH.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) and Binge Eating Disorder (BED) are both characterized by the primary symptoms of binge eating and by significant levels of impairment and psychiatric co-morbidity, affecting approximately 3-5% of the US population. Guided self-help cognitive behavioral (CBT-GSH) therapy has been shown to be an efficacious treatment to reduce binge eating, performing comparatively to full-scale psychotherapy interventions and is a cost-effective empirically supported treatment that has been demonstrated to reduce total health care costs when delivered by trained professionals in primary care settings. Despite the evidence that CBT-GSH offers an effective and financially advantageous treatment for BN and BED, there is evidence of limited uptake for CBT-GSH among both clients and therapists as evidenced by high dropout rates and perceived impediments to therapeutic change. The primary intervention in the CBT-GSH is self-monitoring, which is uniquely effective at reducing binge eating episodes and is packaged with other behavioral strategies including regular eating, using alternatives to binges or purging, problem solving, eliminating rigid dietary practices, and regular weighing. Self-monitoring in CBT-GSH is both time-intensive and cumbersome in its traditional paper format and behavioral strategies require a high degree of engagement outside of session. These burdens lead to reduced therapeutic adherence, which is essential to the efficacy of CBT-GSH. Initial evidence with text messaging interventions suggest increased treatment and self-monitoring adherence for BN. A yet unexplored advantage of mobile application technology is the ability to synthesize real-time data to provide feedback on patient progress. Providing therapists with direct feedback about patient progress has a well-documented effect on treatment outcome and adherence. Thus, mobile application technology offers an innovative opportunity to increase client and therapist uptake of CBT-GSH by (1) reducing the burden of self-monitoring and de-stigmatizing the act of real-time meal recording, (2) offering between-session application of CBT-GSH principles , (3) facilitating feedback to therapists about patient progress. This study proposes to develop a commercial product, the "Noom Monitor," to capitalize on emerging mobile application technology thus enhancing the acceptability and efficacy of CBT-GSH. This will be accomplished by adapting Noom Inc.'s current commercial mobile product, Noom, into a therapy transfer application for individuals with BN. The acceptability, treatment adherence, and preliminary efficacy of the adapted application will be examined through a randomized control trial comparing CBT-GSH + Noom Monitor with traditional CBT-GSH conducted at the Mount Sinai School of Medicine's Eating and Weight Disorders Program. The innovative utilization of technology to assist in mental health interventions has widespread implications outside of this proposal, which will be used to strategize the further development and commercialization of this product.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for DSM-V BN or BED or must have objective binge episodes with sub-threshold BN or BED criteria
* an upper limit BMI of 40
* between the ages of 18 and 55
* are medically stable for outpatient treatment as determined by their primary care physician
* free of psychiatric medications for at least 2-weeks prior to study, or on a stable dose of medication for 4 weeks prior to the study

Exclusion Criteria:

* prior lap band or other bariatric procedure completed
* meeting current of drug or alcohol dependence or bipolar disorder
* active psychotic symptoms by SCID-I screen questions
* current suicidal ideation
* prior Cognitive behavioral therapy for eating disorders
* concurrent psychological treatment of any type
* Previously read Chris Fairburn's Overcoming Binge Eating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination version 16 | up to 9 months
  Frequency of objective binge episodes

SECONDARY OUTCOMES:
Treatment Adherence | 3 months of treatment
  Self-monitoring data from paper and pencil records and smartphone app data

OTHER OUTCOMES:
Acceptability measure assessed by verbal qualitative data | up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hildebrandt, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Hildebrandt T, Michaelides A, Mackinnon D, Greif R, DeBar L, Sysko R. Randomized controlled trial comparing smartphone assisted versus traditional guided self-help for adults with binge eating. Int J Eat Disord. 2017 Nov;50(11):1313-1322. doi: 10.1002/eat.22781. Epub 2017 Sep 27. PMID 28960384